CLINICAL TRIAL: NCT01033994
Title: A Randomized, Double Blind, Placebo-controlled, Multicenter, Single and Multiple Ascending Dose Study of AS902330 (rhFGF-18) Administered Intra-articularly in Patients With Primary Osteoarthritis of the Knee Who Are Not Expected to Require Knee Surgery Within One Year
Brief Title: A Multicenter Study of rhFGF 18 in Patients With Knee Osteoarthritis Not Requiring Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28980
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Fibroblast growth factor 18; Sprifermin
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — fibroblast growth factor 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AS902330 (Experimental)
  Interventions: Biological: AS902330
- Placebo (Placebo Comparator)
  Interventions: Biological: AS902330

INTERVENTIONS:
Biological: AS902330 — 10, 30 or 100 µg intra-articular injection per subject in the Single Ascending Dose (SAD) cohorts and 10, 30 or 100 µg intra-articular injection per week for three weeks per subject in the Multiple Ascending Dose (MAD) cohorts.
  Other Names: rhFGF 18; Recombinant human fibroblast growth factor 18; Sprifermin

SUMMARY:
Osteoarthritis (OA) is one of the most common diseases affecting the joints, usually those that are weight bearing such as the knees. OA is considered to be a disease of the cartilage in the joints even though it involves the whole joint, including the bone and synovium (thin lining of the joints which produces synovial fluid). With time, more and more of the cartilage is destroyed by the disease with inflammation commonly occurring.

AS902330 is expected to increase the production and development of specific bone cells: chondrocytes and osteoblasts (cells that produce and maintain bone and cartilage). This is expected to lead to repair and generation of the cartilage, and a narrowing of the space width between the knee joints in a selected region of the knee cartilage. The purpose of this study is to see how safe treatment with AS902330 is, and to evaluate its effect on the knee cartilage. In addition, the study will also measure the effects of AS902330 in the blood, which reflect disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >= 40 years of age; females must be postmenopausal or surgically sterile
2. Established diagnosis of primary femoro-tibial OA of the target knee by standard American College of Rheumatology Criteria for at least six months (clinical AND radiological criteria)
3. Radiological disease stage 2 or 3 (i.e., clear evidence of OA, but not most advanced disease) in the target knee according to the Kellgren-Lawrence grading of knee OA
4. No major knee surgery (e.g., partial or total knee replacement, interventional arthroscopy) in the target knee planned for at least 12 months after first injection of the study drug
5. Documented need for symptomatic PRN (as needed)-treatment for OA in the target knee with systemic non-steroidal anti-inflammatory drugs (NSAIDs) and/or other analgesics.
6. Total WOMAC score between 24 and 72 (out of 96, corresponding to mild, moderate, or severe, but not extreme OA symptoms) for the target knee while on oral symptomatic treatment at baseline
7. Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
8. Patients must have read and understood the informed consent form, and must have signed it prior to any study-related procedure

Exclusion Criteria:

* any condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation
* clinically significant abnormal hematology (hemoglobin, leucocytes, and platelets), or blood chemistry values (aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), bilirubin, and creatinine
* receipt of any investigational product or any experimental therapeutic procedure within the last 12 weeks preceding screening
* participation in FIH study 27575 or in a different cohort of this study
* i.a. treatment of the target knee with steroids or hyaluronic acid derivatives within the 3 months before baseline
* for MAD cohorts, any contra-indications to MRI according to MRI guidelines
* any condition that would interfere with efficacy or safety assessments in the target knee
* any drug or food supplement with potential disease-modifying effect (glucosamine, diacerin, chondroitin sulfate) unless given at a stable dose over at least 4 weeks prior to first injection
* use of electrotherapy or acupuncture for OA, unless there is a stable regimen for at least 4 weeks before baseline
* any known active infections, including suspicion of intra-articular infection and/or infections that may compromise the immune system such as HIV, Hepatitis B or Hepatitis C infection
* history of sarcoma and/or of other active malignancy within five years, except adequately treated basal cell or squamous cell carcinoma of the skin
* signs and symptoms suggestive of transmissible spongiform encephalopathy
* secondary osteoarthritis: e.g., joint dysplasias, aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos syndrome, Gaucher's disease, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, calcium pyrophosphate deposition disease, or neuropathic arthropathy whatever the cause

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in cartilage thickness in the medial femoro-tibial compartment of the target knee joint, assessed by MRI | 6 and 12 months after first injection
Nature, incidence and severity of local and systemic treatment-emergent adverse events (TEAEs) | MAD Cohorts: 1 year + 1 month; SAD Cohorts: 4 Weeks
Proportion of subjects experiencing AIRs defined as increase of pain by 30mm on a 100mm visual analogue scale (VAS) associated with a self-reported synovial fluid effusion within 3 days following i.a. injection | MAD Cohorts: Week 1, 2, 3, 13 14 and 15 (injections weeks); SAD Cohorts: Week 1
Laboratory assessments, including blood chemistry, hematology, urinalysis, and ECG | MAD Cohorts: Week 0, 4, 13, 17, 52; SAD Cohorts: Weeks 0 & 4

SECONDARY OUTCOMES:
Change in cartilage thickness in the medial femoro-tibial compartment of the target knee joint, assessed by MRI | 52 Weeks
Change in total cartilage volume and thickness in the other compartments of the target knee joint, assessed by MRI | 52 Weeks
Change over time of structural as well as compositional parameters of the knee joint (e.g. cartilage and bone), evaluated by MRI | 52 Weeks
Change in WOMAC (Western Ontario MacMaster Osteoarthritis Questionaire) total score in the target knee from 5-point Likert scales | 52 Weeks
Change in WOMAC Function and Pain index scores in the target knee | 52 Weeks
Change in osteoarthritis (OA) pain in the target knee on a 100mm visual analogue scale (VAS) | 52 Weeks
Change in JSW in the target knee by x-ray | 52 Weeks
Presence of anti-AS902330 antibodies | 52 Weeks
Blood levels of AS902330 | 52 Weeks
MRI at 3 months, score on WOMAC questionnaire at 3, 6 and 12 months. | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Donatus Dreher, MD, PhD, Study Director — Merck Serono S.A., Geneva
Locations (28):
- UMHAT "Sv. Ivan Rilski", Clinical Research Unit for Phase I, Sofia, Bulgaria
- Canada (6):
  - SKDS Research, Inc., Newmarket
  - Kells Medical Research Group, Pointe-Claire
  - Centre de rhumatologie St-Louis, Québec
  - Groupe de Recherche en Maldies Osseuses de Quebec, Québec
  - London Road Diagnostic Clinic, Sarnia
  - Albion Finch Medical Centre, Toronto
- Croatia (3):
  - Clinical hospital Split, Split
  - Clinical Hospital "Sestre Milosrdnice", Zagreb
  - Polyclinic for internal medicine, gynecology, radiology, physical medicine and rehabilitation, Zagreb
- Finland (3):
  - Kuopio University Hospital, Department of Ortopaedics, Kuopio
  - Oulu University Hospital, Surgical and Intensive Care Division, Oulu
  - Turku University Central Hospital, Orthopedic Research Unit, Turku
- PAREXEL International GmbH, Berlin, Germany
- Poland (6):
  - NZOZ Centrum Medyczne Artur Racewicz, Bialystok
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - REUMED Sp. z o.o.,, Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej Nasz Lekarz, Torun
  - Centrum Leczenia Chorob Cywilizacyjnych, Warsaw
  - Centrum Medyczne OSTEOMED Sp. z o.o., Warsaw
- Serbia (3):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute of Rheumatology Resavska 69, Belgrade
  - • Name: Institute of diagnostic, prevention and rechabilitation of cardiovascular and rheumatoid diseases, Niška Banja
- South Africa (3):
  - FARMOVS-PAREXEL (Pty) Ltd, University of the Free State, Bloemfontein
  - PAREXEL -George, George
  - PAREXEL-Port Elizabeth, Mercantile Hospital, Port Elizabeth
- Sweden (2):
  - Ortopediska mottagningen, Hässleholm
  - Kirurg- och ortopedkliniken Kungälvs sjukhus, 442 83 Kungälv, Kungälv

REFERENCES:
- [Result] Lohmander LS, Hellot S, Dreher D, Krantz EF, Kruger DS, Guermazi A, Eckstein F. Intraarticular sprifermin (recombinant human fibroblast growth factor 18) in knee osteoarthritis: a randomized, double-blind, placebo-controlled trial. Arthritis Rheumatol. 2014 Jul;66(7):1820-31. doi: 10.1002/art.38614. PMID 24740822
- [Result] Onuora S. Osteoarthritis: Sprifermin shows cartilage-protective effects in knee OA. Nat Rev Rheumatol. 2014 Jun;10(6):322. doi: 10.1038/nrrheum.2014.68. Epub 2014 May 6. No abstract available. PMID 24798571
- [Derived] Roemer FW, Aydemir A, Lohmander S, Crema MD, Marra MD, Muurahainen N, Felson DT, Eckstein F, Guermazi A. Structural effects of sprifermin in knee osteoarthritis: a post-hoc analysis on cartilage and non-cartilaginous tissue alterations in a randomized controlled trial. BMC Musculoskelet Disord. 2016 Jul 9;17:267. doi: 10.1186/s12891-016-1128-2. PMID 27393009
- [Derived] Eckstein F, Wirth W, Guermazi A, Maschek S, Aydemir A. Brief report: intraarticular sprifermin not only increases cartilage thickness, but also reduces cartilage loss: location-independent post hoc analysis using magnetic resonance imaging. Arthritis Rheumatol. 2015 Nov;67(11):2916-22. doi: 10.1002/art.39265. PMID 26138203